CLINICAL TRIAL: NCT02460263
Title: A Prospective Multicenter, Open Label, Non-Randomized, Cross-Over Study Evaluating the Use of the Tablo Hemodialysis System In-Center and In-Home by Subjects With End Stage Renal Disease (ESRD) Who Are on Stable Dialysis Regimens
Brief Title: The EvAluation of TaBlo In-CLinic and In-HOme
Acronym: TABLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Outset Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2014-01
Record Dates: First submitted 2015-05-20; First posted 2015-06-02 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled in the trial for approximately 21 weeks according to the following schedule:
  * Run-in, In-Center - Subjects undergo study staff administered dialysis treatment 4 times/week for 1 week
  * Treatment Period 1, In-Center - Subjects undergo study staff administered dialysis treatment 4 times/week for 32 treatments (approximately 8 weeks)
  * In-Home Transition - Subjects undergo device training for the study, perform self-care dialysis 4 times/week for approximately 4 weeks, and are assessed for stability in the new care environment.
  * Treatment Period 2, In-Home - Subjects undergo self-care dialysis treatment 4 times/week for 32 treatments (approximately 8 weeks)

ARMS (2):
- In-Center (Placebo Comparator): Staff administered treatments in-center using the device
  Interventions: Device: Tablo Hemodialysis System
- In-Home (Experimental): Patient administered treatments in-home using the device
  Interventions: Device: Tablo Hemodialysis System

INTERVENTIONS:
Device: Tablo Hemodialysis System

SUMMARY:
The purpose of this study is to evaluate the Tablo Hemodialysis System when used In-Center by trained individuals and In-Home by trained Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject has end stage renal disease (ESRD) adequately treated by maintenance dialysis achieving a Kt/V ≥ 1.2 and has been deemed stable for at least three months by his/her treating nephrologist.
* Subject has a well-functioning and stable vascular access that allows a blood flow of at least 300 ml/min.

Exclusion Criteria:

* Life expectancy less than 12 months from first study procedure.
* Subject has had a recent major cardiovascular adverse event within the last 3 months.
* Subject has New York Class III or IV Congestive Heart Failure, or ejection fraction less than 30%.
* Subject with fluid overload due to intractable ascites secondary to liver cirrhosis.
* Subject has uncontrolled blood pressure.
* Subject is intolerant to heparin.
* Subject is seroreactive for Hepatitis B Surface Antigen.
* Subject has an active, life-threatening, rheumatologic disease.
* Subject has a history of adverse reactions to dialyzer membrane material.
* Subject is expected to receive an organ transplant during the course of the study.
* Subject has a life-threatening malignancy actively receiving treatment that would prevent successful completion of the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Outset Medical, San Jose, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 8 dialysis centers throughout the U.S.
Pre-assignment Details: A run-in period of 1 week (4 hemodialysis treatments) was required on the Tablo Hemodialysis System prior to the first period.
Groups:
- In-Center Dialysis, Then In-Home Dialysis: Subjects first entered the In-Center period of the trial before transitioning to the In-Home period. Dialysis treatments were based on physician prescription (clearance and volume targets) and included the following schedules:
  * Treatment Period 1, In-Center - Subjects received study staff administered dialysis treatment 4 times/week for 32 treatments (approximately 8 weeks)
  * In-Home Transition- Subjects received device training and performed self-care dialysis 4 times/week for approximately 4 weeks, and were assessed for stability in the new care environment.
  * Treatment Period 2, In-Home - Subjects received self-care dialysis treatment 4 times/week for 32 treatments (approximately 8 weeks)
Period: In-Center Period
Arm/Group | In-Center Dialysis, Then In-Home Dialysis
Started | 30
Completed | 30
Not Completed | 0
Period: Transition Period
Arm/Group | In-Center Dialysis, Then In-Home Dialysis
Started | 30
Completed | 28
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Period: In-Home Period
Arm/Group | In-Center Dialysis, Then In-Home Dialysis
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intention-To-Treat (ITT) Population: The ITT population was defined as all participants who were enrolled and fulfilled inclusion criteria.
Arm/Group | Intention-To-Treat (ITT) Population
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Vascular Access Type [Count of Participants; unit: Participants]
  Fistula | 23
  Catheter | 4
  Graft | 3

OUTCOME MEASURES:

1. Primary Outcome: Weekly Standardized Dialysis Adequacy
Description: Weekly standardized dialysis adequacy (stdKt/V) was measured using the second-generation formula of Daugirdas. This formula normalizes urea clearance among heterogeneous hemodialysis schedules, where K=dialyzer clearance or urea, t=treatment time, and V=subject's volume of urea distribution. stdKt/V values of ≥ 2.1 are regarded as being adequate.
Time Frame: 8 weeks per period
Population: Intention-to-treat (ITT) population with no imputation of missing values.
Measure: Mean (Standard Deviation); unit: Weekly Standardized Kt/V
Groups:
- In-Center: Staff administered hemodialysis treatments for participants 4 times per week for 8 weeks In-Center using the Tablo system
- In-Home: Participants administered hemodialysis treatments In-Home using the Tablo system
Arm/Group | In-Center | In-Home
Number analyzed (Participants) | 30 | 28
Weekly Standardized Kt/V | 2.8 (0.3) | 2.8 (0.3)

2. Primary Outcome: Incidence of Pre-Specified Adverse Events
Description: All adverse events (AEs) observed in the trial were reviewed by an independent Clinical Events Committee (CEC). AEs adjudicated into the following pre-specified categories were included in the outcome measure:
  1. Serious Adverse Event
  2. Allergic Reaction: to dialyzer, blood tubing or chemical disinfectant.
  3. Blood Loss: that leads to death, transfusion or fluid resuscitation with greater than 1 liter of crystalloid IV fluids.
  4. Hemolytic Reaction: due to disinfectant exposure, dialysate temperature, mechanical failure or other device related causes.
  5. Infection: any infection related to catheter, its tunnel or exit site, AV fistula, or AV graft.
  6. Intra-Dialysis Event: a significant clinical event such as loss of consciousness, cardiac arrest, or seizure caused by device failure.
  7. Vascular Access Complications
  8. Pyrogenic Reaction
Time Frame: 8 weeks per period
Population: Safety Population
Measure: Number; unit: Adverse Events
Groups:
- In-Center: Staff administered hemodialysis treatments for participants In-Center using the Tablo system
Arm/Group | In-Center | In-Home
Number analyzed (Participants) | 30 | 28
Adverse Events | 2 | 6

3. Secondary Outcome: Ultrafiltration Rate Success
Description: The Ultrafiltration (UF) rate was calculated using the following method:
  UF rate = (Fluid Removal Goal + Rinse Back Volume) / Treatment Duration.
  Where: Fluid Removal Goal = (Today's Weight - Prescribed Estimated Dry Weight)
  And: Rinse Back Volume = The volume of saline, 300mL, returned to the patient at the end of treatment.
  Each dialysis treatment was flagged as a success with respect to UF if the actual UF rate was within 10% of the prescribed UF rate. The mean (i.e., success proportion) and standard deviation were computed by treatment period across all subjects, where the denominator for the mean calculations was the total number of treatments in each treatment period for which the subjects contributed non-missing UF data.
Time Frame: 8 weeks per period
Population: Intention-to-treat (ITT) population with no imputation of missing values.
Measure: Number; unit: Percentage of Dialysis Treatments
Arm/Group | In-Center | In-Home
Number analyzed (Participants) | 30 | 28
Percentage of Dialysis Treatments | 94 | 94

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the following time periods: In-Center Period: 8 weeks Transition Period: 4 weeks In-Home Period: 8 weeks
Description: All AEs were required to be reported in the trial and were assessed through participant questionnaires, investigator assessments and laboratory testing.
  AEs were reviewed by an independent Clinical Events Committee (CEC) and adjudicated into two categories:
  1. Pre-specified AEs (e.g., SAEs and/or treatment-related events)
  2. Unrelated to Tablo System
  Unrelated AEs were fully adjudicated for seriousness / relatedness, but were not assigned a specific AE term (MedDRA).
Groups:
- Transition Period: Staff and participant administered hemodialysis treatments using the Tablo system
Arm/Group | In-Center | Transition Period | In-Home
All-Cause Mortality (participants affected / at risk) | 0/30 | 1/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/30 | 2/30 | 2/28
Other Adverse Events (participants affected / at risk) | 14/30 | 6/30 | 10/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-Center (N=30) | Transition Period (N=30) | In-Home (N=28)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (2)
Vascular Access Site Complication (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid Overload (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-Center (N=30) | Transition Period (N=30) | In-Home (N=28)
Unrelated to Tablo System (Investigations) | 13 (16) | 6 (9) | 9 (14) — Adverse events deemed unrelated to Tablo Hemodialysis System
Blood Loss from Dialyzer & Lines (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT02460263/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT02460263/SAP_001.pdf